CLINICAL TRIAL: NCT05082311
Title: Prospective Cohort Study of Objective Cardiac and Vascular Changes in Pheochromocytoma and Paraganglioma and Their Reversal Following Curative Surgery
Brief Title: Cardiac and Vascular Changes in Pheochromocytoma and Paraganglioma
Acronym: PheoCard
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Gaurav Agarwal, Professor of Endocrine Surgery, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2018-185-Mch-EXP-4
Record Dates: First submitted 2021-07-25; First posted 2021-10-18 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Pheochromocytoma; Paraganglioma; Cardiovascular Morbidity
Keywords: Pheochromocytoma; Paraganglioma; Cardio vascular manifestations; Cardiomyopathy; Speckle Tracking echocardiography
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Cardiomyopathies | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Pheochromocytoma/Paraganglioma (secretory, extra adrenal pheochromocytoma): Patients included in this cohort (n=50) are those who are diagnosed of Pheochromocytoma / Paraganglioma, willing to consent for the study and not on α-blockade at the time of recruitment into study, while can be on any other anti hypertensives
  Patients in this group, besides the usual evaluation of Pheochromocytoma / Paraganglioma, will also undergo detailed cardiac and vascular evaluation, which will be done at diagnosis, at 7- 10 days of α-blockade, and 7 days, 3 and 6 months post adrenalectomy/ Paraganglioma excision The cardiovascular evaluation includes 2D-echocardiography, speckle tracking Echo (for measuring global longitudinal strain), serum NT-proBNP estimation and flow mediated vasodilatory studies by Doppler Ultrasonography of the brachial artery to assess the endothelial dependent and smooth muscle dependent vasodilatory responses
  Interventions: Other: Observational study
- Essential Hypertensive Groups: This is a contemporary age- and gender-matched control group This group includes 10 newly detected (within 3 months) Essential Hypertensive patients, who will undergo treatment with standard anti- HT medications Cardiac evaluation will be done at baseline and after 3 months of anti hypertensive medications
  Interventions: Other: Observational study
- Healthy Individuals: This is a contemporary age- and gender-matched control group This group includes 10 Healthy individuals (normal in physical examination, ECG , Echo), that include hospital staff nurses, technicians, doctors whom would be requested to volunteer Cardiac evaluation will be done at the start of study and after 6 months
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This is an observational study

SUMMARY:
PHEOCHROMOCYTOMA (PCC)/ PARAGANGLIOMA are catecholamine secreting tumors with varied manifestations. Besides hypertension, PCC patients may have subclinical to overt cardiac and vascular dysfunction, which are important to recognize to minimize perioperative morbidity and mortality. Cardiovascular (CV) dysfunction can be in the form of hypertension, left ventricular (LV) hypertrophy, heart failure, cardiomyopathy, dysrhythmias, angina and Myocardial infarction. Literature search revealed a few retrospective and a few prospective studies, including one prospective follow up study conducted at SGPGIMS to document CV changes in PCC. Our institutional study was the first to document the nature and extent of CV dysfunction and cardiomyopathy and their reversal after surgical cure. The studies revealed that PCC patients had significantly higher LV mass index, higher LV diastolic dysfunction, subclinical impaired LV systolic function. Earlier studies postulated apparent improvement in various cardiac indices even with selective α-blockade and continued after surgical cure, with near normalization at 3 -6 months postoperatively. Detailed cardiac and vascular evaluation in PCC patients can be of help in preoperative optimization of cardiac risk and may provide prognostic information The literature on PCC-mediated CV dysfunction and catecholamine cardiomyopathy is largely limited to case reports and retrospective studies, with few reports of their reversal after curative PCC operations. Whether the duration of disease influence the function of heart was not apparently addressed in earlier trials. Trials that established the differences in the degree of cardiac dysfunction between normotensive and hypertensive PCC patients involved smaller proportion of study subjects. Sub clinical changes in endomyocardium was presumed but not objectively assessed and hence its reversal after surgical cure is uncertain.

The aim of this research is to study the cardiac and vascular changes in Pheochromocytoma/ Paraganglioma patients and their reversal following curative surgery

DETAILED DESCRIPTION:
The aim of this research is to study the cardiac and vascular changes in Pheochromocytoma/ Paraganglioma patients and their reversal following curative surgery

This prospective, case-control study is conducted at SGPGIMS, Lucknow, India, tertiary care referral institute, between January 2019 and September 2021 after approval from institutional ethics committee. The study group includes 50 biochemically and histopathology proven PCC /Paraganglioma patients, who after 1 to 3 weeks of α-adrenoceptor blockade with oral prazosin undergo primary laparoscopic or open surgery. Cure of hypercatecholaminism will be documented by normal 24-hour urinary fractionated metanephrine values at 7-10 days postoperatively.

Two contemporary age- and gender-matched control groups includes 10 newly detected (withtin 3 months) Essential Hypertensive (E-HT) patients, who will undergo treatment with standard anti- HT medications and 10 Healthy individuals (normal in physical examination, ECG , Echo), that include hospital staff nurses, technicians, doctors whom would be requested to volunteer.

METHODOLOGY

Patients in the study group, besides the usual evaluation of PCC, also undergo detailed cardiac and vascular evaluation, at diagnosis, at 7- 10 days of α-blockade, and 7 days, 3 and 6 months post adrenalectomy/ Paraganglioma excision and in control groups - E-HT controls, cardiac evaluation is done at diagnosis and after 3 months of anti HT medications ; in Healthy individuals, cardiac evaluation is done at the start of study and after 6 months.

The CV evaluation includes 2D-echocardiography, speckle tracking Echo (for measuring global longitudinal strain), serum NT-proBNP estimation and flow mediated vasodilatory studies by Doppler Ultrasonography of the brachial artery to assess the endothelial dependent and smooth muscle dependent vasodilatory responses

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of Pheochromocytoma (PCC) / Paraganglioma (secretory, extra adrenal PCC) Patients willing to consent for the study Patients not on α-blockade at the time of recruitment into study, can be on any other anti hypertensives

Exclusion Criteria:

* Non-secretory Paraganglioma Patients who refuse consent, not compliant in follow up Patients who are on α- blockade already Essential Hypertensives with compounding comorbidities that could interfere with cardio vascular evaluation

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study group will include 50 biochemically and histopathology proven Pheochromocytoma /Paraganglioma patients, who after 1 to 3 weeks of α-adrenoceptor blockade with oral prazosin will undergo primary laparoscopic or open surgery. Cure of hypercatecholaminism will be documented by normal 24-hour urinary fractionated metanephrine values at 7-10 days postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change of Systolic function indices measurement by 2D-Echocardiography from Baseline versus after alpha blockade and after surgery | at baseline (Day 1), at Day 7- 10 after initiation of α-blockade, and 7 days, 3 and 6 months post adrenalectomy/ Paraganglioma excision
  Left ventricle end systolic and end diastolic diameter in millimeter
Change of Systolic function indices measurement by 2D-Echocardiography from baseline versus after alpha blockade and after surgery | at baseline (day 1), at Day 7- 10 after initiation of α-blockade, and 7 days, 3 and 6 months post adrenalectomy/ Paraganglioma excision
  Left ventricle end systolic and end diastolic volume dimensions in milliliter
Change of Systolic function index measurement by 2D-Echocardiography from Baseline at after alpha blockade and at after surgery | at baseline (Day1), at Day 7- 10 after initiation of α-blockade, and 7 days, 3 and 6 months post adrenalectomy/ Paraganglioma excision
  Left ventricle Ejection fraction by Simpsons method in percentage
Change of Diastolic function index measurement by pulsed wave doppler echocardiography from baseline versus after alpha blockade and after surgery | at baseline (Day 1), at Day 7- 10 after initiation of α-blockade, and 7 days, 3 and 6 months after adrenalectomy/ Paraganglioma excision
  Peak velocities of the early (E) and Late phase (A) of the mitral valve inflow pattern and their ratio in centimeter per second
Change of Diastolic function indices measurement by pulsed wave doppler echocardiography from baseline versus after alpha blockade and after surgery | at baseline (day 1), at day 7- 10 after initiation of α-blockade, and 7 days, 3 and 6 months after adrenalectomy/ Paraganglioma excision
  Flow rate across mitral valve in centimeter per second and deceleration time in millisecond
Change in Speckle tracking echocardiographic parameters at Baseline versus after alpha blockade and at after surgery | at baseline (Day 1), at Day 7- 10 after initiation of α-blockade, and 7 days, 3 and 6 months post adrenalectomy/ Paraganglioma excision
  Left ventricle global longitudinal strain in percentage
Change in Speckle tracking echocardiographic parameters from Baseline in comparison to after alpha blockade and after surgery | at baseline (Day 1), at Day 7- 10 after initiation of α-blockade, and 7 days, 3 and 6 months post surgery
  Left ventricle global circumferential strain in percentage
Change in Vascular Function indices by doppler Ultrasonography of the brachial artery from baseline at after alpha blockade and at after surgery | at baseline (Day 1), at Day 7- 10 after initiation of α-blockade, and 7 days, 3 and 6 months post adrenalectomy/ Paraganglioma excision
  Flow mediated dilation of brachial artery diameter pre and post sublingual isosorbide dinitrate in millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Agarwal, MS,DNB,PDC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, India
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Agarwal G, Sadacharan D, Kapoor A, Batra A, Dabadghao P, Chand G, Mishra A, Agarwal A, Verma AK, Mishra SK. Cardiovascular dysfunction and catecholamine cardiomyopathy in pheochromocytoma patients and their reversal following surgical cure: results of a prospective case-control study. Surgery. 2011 Dec;150(6):1202-11. doi: 10.1016/j.surg.2011.09.001. PMID 22136841
- [Result] Agarwal G, Mishra AK, Kapoor A, Agarwal A, Bhatia E, Mishra SK. Reversal of catecholamine induced cardiomyopathy in a patient with bilateral malignant pheochromocytoma. J Assoc Physicians India. 2001 Dec;49:1193-6. PMID 11996444
- [Result] Ding L, Zhu WL, Zeng ZP, Li HZ, Ji J, Fang LG, Sun JP. Subclinical left ventricular systolic dysfunction detected by two-dimensional speckle tracking echocardiography in patients with pheochromocytoma and paraganglioma and preserved ejection fraction. Echocardiography. 2018 Feb;35(2):184-189. doi: 10.1111/echo.13752. Epub 2017 Nov 22. PMID 29168209
- [Derived] Vishvak Chanthar KMM, Khanna R, Agarwal G, Rout SR, Kapoor A, Sabaretnam M, Chand G, Mishra A, Agarwal A, Mishra SK. Cardiac Changes and Their Reversal Following Curative Surgery in Pheochromocytoma: PheoCard Prospective Cohort Study. World J Surg. 2023 Feb;47(2):304-311. doi: 10.1007/s00268-022-06731-6. Epub 2022 Oct 10. PMID 36210362